CLINICAL TRIAL: NCT04820725
Title: The Effects of Postural Changes on Plantar Pressure in Patients With Ankylosing Spondylitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Songul Baglan Yentur, Asistant Professor, Firat University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 05-06
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-01

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis,; posture; plantar pressure
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Gait

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Patients whose BASMI score is 2 will be included in the study
  Interventions: Diagnostic Test: Plantar pressure and gait
- Control group (Experimental): Patients whose BASMI score is 0 and 1 will be included in the study
  Interventions: Diagnostic Test: Plantar pressure and gait

INTERVENTIONS:
Diagnostic Test: Plantar pressure and gait — Gait analyses (cadence, stride length, swing phase duration, step duration and double stand duration) will be evaluated using Win-Track platform (MEDICAPTEURS Technology, France).

SUMMARY:
Ankylosing Spondlitis (AS) is a chronic, rheumatic disease. Foot and ankle involvement may stem from both postural changes in patients seen spinal deformity with the progress of the disease and enthesitis. The purpose of the study is to investigate the relationship plantar pressure distribution and balance, mobility and disease activity in AS patients and to compare AS patients with and without postural changes and healthy subjects.

DETAILED DESCRIPTION:
Ankylosing Spondlitis (AS) is a chronic, rheumatic disease. Reduction in flexibility and mobility is important factors that can cause impairment quality of life, reduction of exercise tolerance and pulmonary capacity with the progression of AS. Extra articular symptoms such as neurologic, cardiovascular and pulmonary involvement affect morbidity and mortality rate. Foot and ankle involvement may stem from both postural changes in patients seen spinal deformity with the progress of the disease and enthesitis. Şahlı et al. concluded that 52% of AS patients had foot involvement but 35% of the patients had symptoms. To be determined plantar pressure distribution is important to be decided body weight distribution, postural control and selection of shoes. The purpose of the study is to investigate the relationship plantar pressure distribution and balance, mobility and disease activity in AS patients and to compare AS patients with and without postural changes and healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are aged between 18-55 years,
* Patients who got diagnosed according to Modified New York criteria
* Patients who are being followed at Firat University Department of Rheumatology.

Exclusion Criteria:

* Patients who have exercise habits
* Incooperation
* Malignancy
* Pregnancy
* Patients who have changes of medical treatment in the last 3 months
* Patients who have another disease that can effect pulmonary functions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10-31 (Estimated); Primary Completion 2022-08-17 (Estimated); Study Completion 2022-12-02 (Estimated)

PRIMARY OUTCOMES:
Gait analyses | 3 minutes
  plantar pressure distribution

SECONDARY OUTCOMES:
Bath Ankylosing Spondylitis Metrology Index | 5 minutes
  Spinal mobility will assessed and scored by Bath Ankylosing Spondylitis Metrology Index (BASMI). There are five measurements including lateral lumbar flexion, tragus-to-wall distance, lumbar flexion (Modified Schober), maximal intermalleolar distance and cervical rotation according to the index. Each subscale is scored between 0 and 10. All points are then averaged to calculate total score. Higher values represent worse outcomes.
Bath Ankylosing Spondylitis Disease Activity Index | 1 minute
  Bath Ankylosing Spondylitis Disease Activity Index which consists of 6 questions will be used to evaluate disease activity. BASDAI is a composite index, consisting of an assessment on a 10 cm horizontal visual analog scale of fatigue, axial pain, peripheral pain, enthesopathy and stiffness. Fifth and sixth questions are averaged. Addition to this score, other questions are averaged. Total score is between 0 and 10. Higher score represent worse outcome.
Time up and go test | 1 minute
  The patient starts in a seated position. The patient stands up upon therapist's command: walks 3 meters, turns around, walks back to the chair and sits down. The time stops when the patient is seated.

CONTACTS AND LOCATIONS:
Overall Officials: Süleyman S Koca, Study Director — Firat University
Locations (1):
- Songul Baglan Yentur, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sahli H, Bachali A, Tekaya R, Mahmoud I, Sedki Y, Saidane O, Abdelmoula L. Involvement of foot in patients with spondyloarthritis: Prevalence and clinical features. Foot Ankle Surg. 2019 Apr;25(2):226-230. doi: 10.1016/j.fas.2017.10.016. Epub 2017 Nov 10. PMID 29409278
- [Background] Aydin E, Turan Y, Tastaban E, Kurt Omurlu I, Sendur OF. Plantar pressure distribution in patients with ankylosing spondylitis. Clin Biomech (Bristol). 2015 Mar;30(3):238-42. doi: 10.1016/j.clinbiomech.2015.02.003. Epub 2015 Feb 8. PMID 25684149